CLINICAL TRIAL: NCT04270669
Title: A Nonrandomized, Open-label Study to Evaluate the Safety and Pharmacokinetics of Multiple Administration of RC28-E Injection (a Chimeric Decoy Receptor Trap Fusion Protein by Dual Blockage of VEGF and FGF-2) in Subjects With Wet Age-Related Macular Degeneration
Brief Title: Evaluation of RC28-E Injection in Wet Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28C001
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Wet Age-Related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RC28-E 0.5mg (Experimental): In the loading phase (from week 0 to week 8), the study eye will receive intravitreal injection of 0.5mg RC28-E every 4 weeks, for 3 consecutive times; In the PRN phase (from week 12 to week 48), the study eye will receive the same dose on an as needed (PRN) schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: intravitreal injection of RC28-E 0.5mg
- RC28-E 1.0mg (Experimental): In the loading phase (from week 0 to week 8), the study eye will receive intravitreal injection of 1.0 mg RC28-E every 4 weeks, for 3 consecutive times; In the PRN phase (from week 12 to week 48), the study eye will receive the same dose on an as needed (PRN) schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: intravitreal injection of RC28-E 1.0mg
- RC28-E 2.0mg (Experimental): In the loading phase (from week 0 to week 8), the study eye will receive intravitreal injection of 2.0 mg RC28-E every 4 weeks, for 3 consecutive times; In the PRN phase (from week 12 to week 48), the study eye will receive the same dose on an as needed (PRN) schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: intravitreal injection of RC28-E2.0mg

INTERVENTIONS:
Biological: intravitreal injection of RC28-E 0.5mg — The patient received one treatment of RC28-E 0.5mg in the test group
  Arms: RC28-E 0.5mg
Biological: intravitreal injection of RC28-E 1.0mg — The patient received one treatment of RC28-E 1.0mg in the test group
  Arms: RC28-E 1.0mg
Biological: intravitreal injection of RC28-E2.0mg — The patient received one treatment of RC28-E 2.0mg in the test group
  Arms: RC28-E 2.0mg

SUMMARY:
This is a non-randomized, open-label, multicenter, 48-week study to investigate the efficacy, safety and pharmacokinetics of RC28-E injection in the treatment of patients with wet age-related macular degeneration by multiple administration.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet the following criteria to be eligible for inclusion in the study:

1. Sign the consent form, willing and able to comply with clinic visits and study-related procedures;
2. Be diagnosed as wet age-related macular degeneration, choroid neovascularization (CNV) in the macular, the study eye is not treated or accepted any treatment 3 months prior to the baseline period, and still had active lesions with a diagnostic criteria according to the 2013 edition of Clinical pathway of age-related macular degeneration in China, the active CNV conforms to any item can be in the following three: New bleeding; OCT shows intraretinal fluid or subretinal fluid; Fundus angiography revealed fluorescein leakage;
3. Aged 50 years to 80 years, male or female;
4. BCVA ETDRS letters score of 73 to 34 in the study eye.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. The study eye had vitreous hemorrhage within 2 months before screening;
2. The study eye had scars or atrophy involving the fovea which indicating severe irreversible visual impairment;
3. The study eye had significant refractive media opacity, including cataract, may interfere with visual assessment;;
4. The study eye had pseudoexfoliation syndrome, central retinal vein occlusion, intraocular hemorrhage resulting in decreased vision, rhegmatogenous retinal detachment, macular hole, choroidal neovascularization (CNV) for any reason other than wAMD (such as vascular striation, ocular histoplasmosis, pathological myopia, trauma, etc.);
5. The study eye had subretinal or intra-retinal bleeding with bleeding area ≥ 50% of the total lesion area, or subfoveal bleeding with bleeding area was ≥4 optic disc areas;
6. The study eye had significant afferent pupillary defect;
7. The study eye was aphakia (excluding artificial lens);
8. The study eye was treated with local/grid laser photocoagulation in macular within 3 months prior to baseline;
9. The study eye had received the following intraocular surgery or laser treatment in macular (such as macular transposition, glaucoma filtrating surgery, transpupillary thermotherapy, vitrectomy, optic neurotomy, etc.); However, subjects which had received verteporfin-photodynamic therapy, cataract surgery, and neodymium yttrium aluminum garnet (YAG) capsulotomy in the study eye more than 3 months prior to baseline is eligible for inclusion;
10. Intraocular pressure in the study eye was≥25mmHg despite medication treatment;
11. Either eye had active ocular infection/inflammation during the screening period, such as conjunctivitis, keratitis, scleritis, blepharitis, endophthalmitis and uveitis;
12. The visual acuity of any eye is less than 19 letters (by ETDRS chart);
13. Either eye or systemic had received anti-angiogenic therapy within 3 months prior to baseline visit (e.g. aflibercept, ranibizumab, conbercept, etc.);
14. Either eye that received IVT corticosteroids (e.g. triamcinolone acetonide, dexamethasone) within 6 months prior to baseline visit or received periocular injection of corticosteroids within 1 month prior to screening;
15. Allergy to sodium fluorescein, indocyanine green, therapeutic or diagnostic protein products, and allergic ≥2 drugs and/or non-drug factors;
16. Uncontrolled diabetes mellitus (HbA1c ≥7%) and/or diabetic patients with diabetic retinopathy;
17. Uncontrolled hypertension (defined as those who received the best treatment regimen, > 180mmHg systolic was measured once, > 160mmHg systolic or > 100mmHg diastolic was measured twice in succession);
18. History of cardiovascular and cerebrovascular events within 6 months of screening visit: myocardial infarction, unstable angina pectoris, ventricular arrhythmias, New York heart association grade II + heart failure, stroke, etc.;
19. History of surgery within 1 month before screening, or have unhealed wounds, fractures, etc.;
20. Uncontrolled clinical disease (such as malignant tumors, severe psychiatric, neurological, cardiovascular, respiratory disease or other systemic diseases);
21. Platelets count ≤100×10^9/L, thrombin time and prothrombin time exceeding more than 3 second above the upper limit of the normal range (The normal range of the clinical trial institution was taken as the standard); with active disseminated intravascular coagulation or significant bleeding tendency prior to screening; using anticoagulants or antiplatelet aggregation drugs in addition to aspirin/NASIDs within 14 days before screening;
22. Pregnant or lactating women. Subjects of child-bearing age (male and female) do not agree to use effective contraception (such as intrauterine devices, acyeterion or condoms) throughout the study period and 30 days after the end of the visit;
23. Those who participated in clinical trials for 3 months or 5 half-lives of the investigational product (the longer the time) before the baseline period;
24. Those who considered unsuitable for enrollment by investigator.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Mean change of BCVA from baseline at 12 week; | Baseline, Week 12
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Mean change of BCVA from baseline at 48 week; | Baseline, Week 48
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Incidence and severity of AEs | Baseline up to Week 48
  To evaluate the safety of multiple intravitreal injection of RC28-E of each group.）

SECONDARY OUTCOMES:
The pharmacokinetic (PK) characteristics of RC28-E; | Baseline up to Week 48
  Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method. These data were analyzed using a noncompartmental pharmacokinetic (PK) method.
Frequency of administration RC28-E within 48 weeks; | Baseline up to Week 48
  Number of intravitreal injections
Mean change of BCVA from baseline at Protocol Specified Time-Points. | Baseline up to Week 48
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China